CLINICAL TRIAL: NCT06571786
Title: Subharmonic Aided Pressure Estimation (SHAPE) for Intracranial Pressure (ICP) Assessment
Brief Title: SHAPE for ICP Assessment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Flemming Forsberg, Professor, Thomas Jefferson University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-2116
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-08

CONDITIONS: Lumbar Puncture
MeSH Terms: interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SHAPE for ICP diagnosis (Experimental)
  Interventions: Drug: Perflutren lipid microsphere

INTERVENTIONS:
Drug: Perflutren lipid microsphere — Definity (Lantheus Medical Imaging, N Billerica, MA) in 25 mL of saline infused for up to 6 minutes
  Other Names: Definity

SUMMARY:
The Subharmonic Aided Pressure Estimation (SHAPE) technique is a noninvasive ultrasound-based imaging technique that can estimate ambient pressure using subharmonic emissions from ultrasound contrast agents. Ultrasound contrast agents are encapsulated microbubbles (mean diameter < 8 µm) with a lipid, protein, or polymer shell that traverse the entire vasculature. When the contrast microbubbles are insonated with relatively high acoustic pressures (>100-150 kPa), these microbubbles act as nonlinear oscillators yielding energy components in the received echo signals at frequencies ranging from the subharmonic (half of transmit frequency) to higher harmonics and even ultraharmonics. Based on empirical evidence, the subharmonic signal exhibits a sigmoidal relationship with incident acoustic pressure i.e., subharmonic signal can be divided into occurrence, growth and saturation stages. In the growth stage, the subharmonic signal has shown sensitivity to ambient pressure characterized by an inverse linear relationship between subharmonic signal and ambient pressure changes. This inverse linear relationship forms the basis for the SHAPE technique. Several pre-clinical and clinical studies have been conducted to utilize the SHAPE technique for in vivo pressure estimation e.g., to diagnose portal hypertension, to estimate intra-cardiac pressures and to determine interstitial fluid pressures. The core imaging mode underpinning the SHAPE technology (subharmonic imaging) is now available on some commercial scanners. In the proposed pilot study, the SHAPE technique will be leveraged for monitoring intracranial pressure (ICP). The use of SHAPE technique for the ophthalmic artery could potentially provide an accurate noninvasive method of measuring ICP in patients with idiopathic intracranial hypertension (IIH) and other conditions of raised ICP, which would revolutionize the field.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for lumbar puncture to assess ICP pressures
* Age over 18.

Exclusion Criteria:

* Pregnant or nursing
* Medically unstable
* Allergy to any components of Definity.
* Unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Comparing SHAPE to lumbar puncture pressure measurements | 1 year
  Use of the SHAPE technique for measuring ophthalmic artery pressure in patients undergoing lumbar puncture for suspected idiopathic intracranial hypertension and compare the SHAPE data with pressures obtained using lumbar puncture (reference standard)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data generated and/or analyzed during this study are available from the PI upon request.
Supporting Information: Study Protocol, Analytic Code
Time Frame: 12 months after completion of the study